CLINICAL TRIAL: NCT06786845
Title: How is the Pain Experience in Fibromyalgia Affected by the Treatment of Comorbid, Newly Diagnosed Sleep Disorder? a Longitudinal Study (HOPES)
Brief Title: Fibromyalgia and Sleep Disorder Treatment
Acronym: HOPES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOPES
Record Dates: First submitted 2024-11-19; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia; Sleep Disorder
Keywords: Inflammation
MeSH Terms: conditions — Fibromyalgia; Sleep Wake Disorders; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment lege artis (Other): Recruited individuals in the cohort undergoe adequate treatment of the sleep disorder initiated by the sleep specialist at the sleep clinic, and when subjects are considered well treated, the sleep investigation is repeated in connection with follow-up 2-4 months later. Sleep duration and physical activity are measured with an actigraph for 10 days after the first visit when sleep treatment was initiated and 10 days before the follow-up, when the sleep intervention is complete.
  Treatment of sleep disorders is carried out according to lege artis at the sleep clinic at the Pain Center (obstructive sleep apnea syndrome, snoring, restless legs syndrom and periodic limb movements, circadian rhythm disorders, insomnia) and examination of pain intensity before (as part of the FINE study) and after treatment is carried out with pain assessment (quantitatory sensory testing and conditioned pain modulation as well as a new panel with inflammatory markers and lumbal puncture).
  Interventions: Other: Treatment lege artis

INTERVENTIONS:
Other: Treatment lege artis — Adequate treatment of sleep disorders at Sleep clinic

SUMMARY:
This longitudinal study will investigate impact of improved sleep quality on chronic pain, fibromyalgia and how the disrupted sleep pattern alters the neuroenvironment.

DETAILED DESCRIPTION:
The main aim of this study is to evaluate the interaction between pain and sleep, both directly by comparing outcome measures of pain and sleep, and out of one inflammatory perspective using proteomics analyzes. Currently, there is a need for studies that highlight both the above-mentioned interaction and how the inflammatory response in the central nervous system as well as in the systemic circulation is involved. The cohort in existing study (FINE study) is already being used to find associations between these, but as it is a cross-sectional study, the design cannot determinate the causality. The implementation of a longitudinal study where sleep is the single parameter that is modified would add an invaluable scientific basis for the assessment of this complex interplay. Because FINE study also has measurements of both systemic as central immunoactivity, the scientific value becomes very high, and can potentially be helpfull in understanding what happens to pain when sleep is affected, and which immune mediators that are relevant in that dynamic. If it turns out that the treatment of sleep disorders is effective from a pain perspective, it would in addition bring a whole new line of treatment options in fibromyalgia, and emphasize the importance of implementation a proper sleep analysis in the investigation phase for this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia according to 1990 and 2016 ACR (American College of Rheumatology criteria)
* Included in FINE study
* Sleep disorder

Exclusion Criteria:

* Other autoimmune or neuroinflammatory diseases than FM.
* Other dominating pain conditions other than FM (e.g., severe pain due to osteoarthritis, disc herniations etc).
* Severe somatic or psychiatric diseases that would preclude participation or influence results (e.g., cancer, infectious diseases etc).
* Pregnancy.
* Inability to speak and understand Swedish.
* Treatment with anticoagulants.
* High intracranial pressure.
* Ongoing infections.
* Hemophilia.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants
Enrollment: 60 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-09-04 (Estimated); Study Completion 2027-04-12 (Estimated)

PRIMARY OUTCOMES:
Changes in sleep quality | 4 months
  Change in subjective sleep disturbance measured by Pittsburgh Sleep Quality Index, a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. Every item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Change in pain intensity after adequate treatment of sleep disorder | 4 months
  measured by Visual Analog Scale, total scores range from 0 to 10 - with a higher score indicating more severe pain (VAS 0 no pain - VAS 10 severe pain)
Change in daytime sleepiness | 4 months
  Change in sleepiness measured by Epworth Sleepiness Scale, a self-administered questionnaire with 8 questions. Rate, on a 4-point scale (0-3), rik of falling asleep while engaging in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher daytime speepiness.
Change in objective sleep disturbance | 4 months
  Change in objective sleep disturbance measured by 1-night ambulatory polysomnography. A polysomnogram is the gold standard test to help diagnose sleep disorders. It involves measuring brain wave activity, eye, and limb movements whilst monitoring the breathing pattern and pulse rate during sleep. It is a non-invasive test which requires several sensors and electrodes to be placed on specific points of the body.

SECONDARY OUTCOMES:
Change in disease burden | 4 months
  Change in disease burden measured by Fibromyalgia Impact Questionnaire, a brief 10-item, self-administered instrument that measures physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well being. A higher score indicates a greater impact of the syndrome on the person. Each of the 10 items has a maximum possible score of 10. The maximum possible score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Romana Stehlik, PhD, Principal Investigator — Pain center
Locations (1):
- Pain center, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol
Time Frame: Q2 2025 - Q2 2027
Access Criteria: Analyses data - SPSS. Data sharing agreement must be signed and PI will review the review requests